CLINICAL TRIAL: NCT00330044
Title: A Phase I Study of Premetrexed (Alimta) and Carboplatin and Radiation Therapy in Patients With Inoperable Non Small Cell Lung Cancer.
Brief Title: Alimta, Carboplatin and Radiation Therapy for Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05C.276; 2005-19 (Other: CCRRC); JT 1070 (Other: JeffTrial Number)
Record Dates: First submitted 2006-05-24; First posted 2006-05-25 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Inoperable Non Small Cell Lung Cancer
MeSH Terms: interventions — Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Drug (Experimental): Carboplatin and Pemetrexed
  Interventions: Drug: Premetrexed (Alimta); Drug: Carboplatin

INTERVENTIONS:
Drug: Premetrexed (Alimta)
Drug: Carboplatin

SUMMARY:
To determine the safety of Alimta when used with chemoradiation in inoperable non small cell lung cancer

DETAILED DESCRIPTION:
To determine the maximal tolerated dose (MTD) and toxicities of Pemetrexed (Alimta) when administered concurrently with carboplatin and thoracic radiation therapy.

To determine, qualitatively, the occurrence of local tumor responses identified with this regimen.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable Stage II, IIIB or IV non small cell lung cancer. Evaluable disease on planning CT scan Zubrod 0-1 Weight loss equal to or less than 10% 3 months prior to diagnosis FEV1 greater than 1000cc Adequate hematologic, renal and hepatic functions

Exclusion Criteria:

* Small cell cancer Stage I non small cell cancer Prior chemotherapy or thoracic or lower neck radiatio therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-04; Primary Completion 2009-08 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Response and Progression Free Survival | Up to five years after study completion

CONTACTS AND LOCATIONS:
Overall Officials: Maria Werner-Wasik, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University — http://www.kimmelcancercenter.org
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/